CLINICAL TRIAL: NCT01307930
Title: Population Pharmacokinetic Analysis of Anidulafungin in Normal, Overweight and Obese Volunteers
Brief Title: Effect of Weight and/or Obesity on Anidulafungin Drug Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ron Hall, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A10-3616; 5UL1RR024982-02 (NIH)
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Mycoses
Keywords: Echinocandin; Obesity; Pharmacokinetics; Pharmacodynamics; Fungal infection
MeSH Terms: conditions — Obesity; Mycoses | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anidulafungin (Experimental): Six volunteers will have a body mass index (BMI) less than 25 kg/m2, 6 will have a BMI 25-40 kg/m2, and 6 will have a BMI greater than 40 kg/m2.
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — Anidulafungin 100 mg IV (each volunteer will only receive one dose of the study drug)
  Other Names: Eraxis

SUMMARY:
This study will find how weight affects the dosing of a drug called anidulafungin. Currently, the amount of anidulafungin a patient receives is the same regardless of the patient's weight. BMI groups were for enrollment purposes only and not used for ordinal data analysis.

DETAILED DESCRIPTION:
This study is designed to measure drug concentrations in the blood of volunteers administered a single intravenous dose of anidulafungin. The volunteers to be enrolled will not have either candidiasis or any other fungal infection. This is a single center study. Up to a total of 35 adult volunteers will be consented for the study at the Clinical and Translational Research Center (CTRC). Eighteen of these volunteers are needed to complete the study. The others will likely be screen failures, which is more likely in the BMI > 40 kg/m2 group. Volunteers will be admitted to the CTRC for an overnight stay. Half will be female and half male. Six volunteers will have a body mass index (BMI) less than 25 kg/m2, six will have a BMI 25-40 kg/m2, and six will have a BMI greater than 40 kg/m2.

** BMI groups will only be used for patient enrollment and not for data analysis. total body weight will be used as a continuous variable for data analysis. **

Volunteers will have height and weight measured after they have consented to participate. All volunteers in each category will receive a single dose of intravenous anidulafungin of 100 mg. The volunteers will have blood drawn via an intravenous catheter just prior to the dose, and then at 1.5, 8, 16, and 24h after the drug dose. The intravenous catheter is then removed after the 24h blood draw, and the volunteer discharged from the study. The volunteer will be asked to return to the CTRC outpatient center at 48 and 72 hours to have the final 2 blood draws conducted. Subjects who are excluded from study participation due to their laboratory results will be provided with a copy of their results and an explanation of the reason for ineligibility.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age > 18 years old, of all racial and ethnic origins.
* Non-English-speaking Spanish speakers will be included in the study.
* The investigators are recruiting six normal or underweight (BMI < 25 kg/m2), six overweight or obese (BMI 25-40 kg/m2), and six extremely obese (BMI > 40 kg/m2) for this study. This index is calculated using the volunteer's height and weight (Formula: weight (lb) / [height (in)]2 x 703). Half of each group will be male; the other half will be female.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of anidulafungin on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of anidulafungin, so that the pregnancy and postpartum state would be a confounding variable.
* Abnormal liver function tests: transaminases > 3 times upper limit of normal, Alkaline phosphatase > 3 times upper limit of normal, total bilirubin > 3 times upper limit of normal.
* History of allergies to echinocandins.
* Echinocandins are contraindicated for any reason.
* Volunteers unwilling to comply with study procedures.
* Suspected or documented systemic fungal infection.
* Concomitant use of rifamycins, tacrolimus, or cyclosporine.
* Current participation or previous participation within 28 days of enrollment in another research study that involves the use of medication, contrast, or any other compound that may alter blood count and/or blood chemistry (liver function, kidney function or electrolyte balance) (Unless waved by PI).
* Donation of 450mL (one unit) of blood or more within 8 weeks (56 days) prior to study enrollment (Unless waved by PI).
* Creatinine Clearance < 70 ml/min as estimated by the Cockcroft-Gault equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hall, PharmD, MSCS, Principal Investigator — Texas Tech UHSC
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: The study will have 18 participants complete the 72 hour sampling period. Six volunteers will have a body mass index (BMI) less than 25 kg/m2, 6 will have a BMI 25-40 kg/m2, and 6 will have a BMI greater than 40 kg/m2.
  Anidulafungin: Anidulafungin 100 mg IV (each volunteer will only receive one dose of the study drug)
Period: Overall Study
Arm/Group | Anidulafungin
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Serum Clearance of Anidulafungin
Description: How quickly the body eliminates anidulafungin after a single dose
Time Frame: 0-72 hours
Population: Noncompartmental analysis of anidulafungin clearance
Measure: Median (Full Range); unit: L/hr
Groups:
- Anidulafungin: Single dose of 100 mg by IV infusion.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 18
L/hr | 0.94 [0.72 to 1.93]

ADVERSE EVENTS:
Time Frame: 3 days
Description: Adverse events were collected upon report of the participant to study staff.
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anidulafungin (N=20)
Rash (Immune system disorders) | 2 (2) — Event 1: Numbness near lips, SOB, itchiness, diffuse rash near arms and chest, wheezing (not life threatening, resolved with benadryl) Event 2: Infusion, facial numbness with bright red flushing rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No